CLINICAL TRIAL: NCT05993585
Title: The Effects of Cardiac Resynchronisation Therapy on the Frank Starling Mechanism in Patients With Heart Failure
Brief Title: The Effect of CRT on the Frank Starling Mechanism
Acronym: CRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 318500
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pacemaker; Heartfailure
Keywords: Frank Starling Mechanism; CRT

STUDY DESIGN:
Intervention Model Description: Single centre trial - observational cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT Group (Experimental): CRT group: We will include patients with symptomatic heart failure (LV ejection fraction <35% on TTE, NYHA II-IV) and an RV pacing percentage of >40%, thus meeting ESC Criteria for CRT upgrade.
  Interventions: Other: Test Of The Frank Starling Mechanism - Adjustment Of Av Delay And Measurement Of Pre-load -Control
- Control Group (Active Comparator): Control group: patients with an existing dual chamber pacemaker and with preserved ejection fraction
  Interventions: Other: Other: Test Of The Frank Starling Mechanism - Adjustment Of Av Delay And Measurement Of Pre-load -CRT

INTERVENTIONS:
Other: Test Of The Frank Starling Mechanism - Adjustment Of Av Delay And Measurement Of Pre-load -Control — (Control Group): One test of the Starling mechanism Visit 1: Sign consent form, doctor assessment, electrocardiogram (ECG), Starling Test. If patients are in this category, this will be their only research visit
  Arms: CRT Group
Other: Other: Test Of The Frank Starling Mechanism - Adjustment Of Av Delay And Measurement Of Pre-load -CRT — (CRT Group): Two tests of the Starling mechanisms Visit 1: Sign consent form, assessment by doctor, electrocardiogram (ECG), Test of the Starling mechanism Visit 2: CRT upgrade procedure - your Cardiologist will explain this procedure to you. Visit 3: CRT pacing check at 6 weeks post-procedure Visit 4: Assessment by doctor, ECG, Echocardiogram, Test of the Starling mechanism at 6 months post-procedure.
  Arms: Control Group

SUMMARY:
The investigators are examining a scientific principle called the Frank Starling Mechanism and how it relates to Cardiac Resynchronisation Therapy (CRT), a form of pacemaker therapy used in the treatment of heart failure.

The Frank Starling Mechanism is an established biological principle. The law states that the stroke volume of the heart increases in response to an increase in the volume of blood in the ventricles, before contraction, when all other factors remain constant. In other words, the law states that the more blood enters the heart, the more blood is pumped out of the heart with any given beat.

There is some evidence that in some patients with chronic heart conditions, the Frank Starling Mechanism is LESS EFFECTIVE, meaning that the heart is less able to cope with a reduction in heart pumping function over time. There is also evidence that treatment with CRT may IMPROVE the Frank Starling Mechanism - evidence for this has been shown in dog and mice hearts, however, has never been shown in humans.

The investigators aim to conduct a study where subjects undergo an ultrasound scan of the heart (echocardiogram) whilst the participants pacemaker settings are temporarily changed. This allows the investigators to measure the pumping function of the heart as more blood enters the heart. The investigators will perform this test on 20 participants before and after CRT, as well as 20 participants who have pacemakers, but no heart failure. This study aims to test 3 hypotheses.

1. In participants with pacemakers, a REDUCED Frank Starling Mechanism predicts which participants go on to develop heart failure.
2. Treatment with CRT IMPROVES the Frank Starling Mechanism in participants with pacemakers and heart failure.
3. The degree of improvement of the Frank Starling Mechanism after treatment with CRT predicts which participants will respond to this treatment.

DETAILED DESCRIPTION:
The primary research investigation in this study is a non-invasive test of the Frank Starling mechanism, which involves performing a transthoracic echocardiogram (ultrasound scan of the heart) whilst temporarily changing pacemaker settings to mimic conditions such as faster heart rates or increased blood flow to the heart. Measurements taken from the echocardiogram during these changes in pacemaker settings will be used to determine the effectiveness of the heart's Starling Mechanism. This test will last between 20-40 minutes. No special preparation is needed and participants will be able to go home immediately afterwards. Pacemaker settings will be returned to normal once the test is completed.

ELIGIBILITY:
Inclusion Criteria:

* • Ability to provide informed consent to participate and willing to comply with the clinical investigation plan and follow-up schedule.

  * Existing dual chamber pacemaker or ICD including atrial lead and RV lead.
  * RV pacing percentage >40%.
  * CRT group - Severe left ventricular systolic impairment (LVEF≤35%). Clinical symptoms of heart failure despite optimum medical therapy (NYHA class II-IV).
  * Control group - LVEF >50%.

Exclusion Criteria:

* • Previous treated with CRT (existing LV lead/His-Bundle lead/Left Bundle Branch Area lead).

  * Persistent atrial fibrillation
  * Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
  * Participation in other studies with active treatment / investigational arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Difference in starling mechanism | Prior to pacing test (starling mechanism test) and after six months
  1. Difference in maximum change in stroke volume (SV) in millilitres with AV delay modification "Starling mechanics" pre-CRT versus post-CRT (difference between lowest and highest SV).

SECONDARY OUTCOMES:
Left ventricular end-systolic volume (ml) | Prior to pacing test (starling mechanism test) and after six months
  Difference in left ventricular end-systolic volume in millimetres recorded on echocardiogram
Left ventricular ejection fraction (%) | Prior to pacing test (starling mechanism test) and after six months
  Difference in Left ventricular ejection fraction in percent measured on echocardiogram
Quality of life with heart failure symptoms | Prior to pacing test (starling mechanism test) and after six months
  Quality of life in heart failure assessed by Minnesota Living with Heart Failure Questionnaire
Heart failure symptoms | Prior to pacing test (starling mechanism test) and after six months
  New York Heart Association ( NYHA) class - breathlessness on different levels of exercise - from walking on the flat (NYHA 2) up to limited by breathlessness on little movement (NYHA 4)
Packer's clinical composite score | Prior to pacing test (starling mechanism test) and at six months
  Difference in patient outcome measured by the clinical composite score - the score ranges from improved to unchanged or worsened
Difference in baseline Starling mechanics between CRT group and control group | Prior to pacing test (starling mechanism test) and at six months
  Difference in stroke volume in millilitres during the pacing test (starling mechanism test) between the CRT and control group

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Aldo Rinaldi/Professor, MD, FHRS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Steven Niederer/Professor, PhD, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable data will be shared upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Non-identifiable data will only be available after the end of the study
Access Criteria: Fully anonymised data available upon request via email

REFERENCES:
- [Background] Kim JH, Kang KW, Chin JY, Kim TS, Park JH, Choi YJ. Major determinant of the occurrence of pacing-induced cardiomyopathy in complete atrioventricular block: a multicentre, retrospective analysis over a 15-year period in South Korea. BMJ Open. 2018 Feb 8;8(2):e019048. doi: 10.1136/bmjopen-2017-019048. PMID 29439074
- [Background] Curtis AB, Worley SJ, Adamson PB, Chung ES, Niazi I, Sherfesee L, Shinn T, Sutton MS; Biventricular versus Right Ventricular Pacing in Heart Failure Patients with Atrioventricular Block (BLOCK HF) Trial Investigators. Biventricular pacing for atrioventricular block and systolic dysfunction. N Engl J Med. 2013 Apr 25;368(17):1585-93. doi: 10.1056/NEJMoa1210356. PMID 23614585
- [Background] Tayal B, Fruelund P, Sogaard P, Riahi S, Polcwiartek C, Atwater BD, Gislason G, Risum N, Torp-Pedersen C, Kober L, Kragholm KH. Incidence of heart failure after pacemaker implantation: a nationwide Danish Registry-based follow-up study. Eur Heart J. 2019 Nov 21;40(44):3641-3648. doi: 10.1093/eurheartj/ehz584. PMID 31504437
- [Background] Chan JY, Fang F, Zhang Q, Fung JW, Razali O, Azlan H, Lam KH, Chan HC, Yu CM. Biventricular pacing is superior to right ventricular pacing in bradycardia patients with preserved systolic function: 2-year results of the PACE trial. Eur Heart J. 2011 Oct;32(20):2533-40. doi: 10.1093/eurheartj/ehr336. Epub 2011 Aug 29. PMID 21875860
- [Background] Kiehl EL, Makki T, Kumar R, Gumber D, Kwon DH, Rickard JW, Kanj M, Wazni OM, Saliba WI, Varma N, Wilkoff BL, Cantillon DJ. Incidence and predictors of right ventricular pacing-induced cardiomyopathy in patients with complete atrioventricular block and preserved left ventricular systolic function. Heart Rhythm. 2016 Dec;13(12):2272-2278. doi: 10.1016/j.hrthm.2016.09.027. PMID 27855853
- [Background] Ebert M, Jander N, Minners J, Blum T, Doering M, Bollmann A, Hindricks G, Arentz T, Kalusche D, Richter S. Long-Term Impact of Right Ventricular Pacing on Left Ventricular Systolic Function in Pacemaker Recipients With Preserved Ejection Fraction: Results From a Large Single-Center Registry. J Am Heart Assoc. 2016 Jul 21;5(7):e003485. doi: 10.1161/JAHA.116.003485. PMID 27444509
- [Background] Kirk JA, Holewinski RJ, Kooij V, Agnetti G, Tunin RS, Witayavanitkul N, de Tombe PP, Gao WD, Van Eyk J, Kass DA. Cardiac resynchronization sensitizes the sarcomere to calcium by reactivating GSK-3beta. J Clin Invest. 2014 Jan;124(1):129-38. doi: 10.1172/JCI69253. PMID 24292707
- [Background] Stachowski-Doll MJ, Papadaki M, Martin TG, Ma W, Gong HM, Shao S, Shen S, Muntu NA, Kumar M, Perez E, Martin JL, Moravec CS, Sadayappan S, Campbell SG, Irving T, Kirk JA. GSK-3beta Localizes to the Cardiac Z-Disc to Maintain Length Dependent Activation. Circ Res. 2022 Mar 18;130(6):871-886. doi: 10.1161/CIRCRESAHA.121.319491. Epub 2022 Feb 16. PMID 35168370
- [Background] Niederer SA, Plank G, Chinchapatnam P, Ginks M, Lamata P, Rhode KS, Rinaldi CA, Razavi R, Smith NP. Length-dependent tension in the failing heart and the efficacy of cardiac resynchronization therapy. Cardiovasc Res. 2011 Feb 1;89(2):336-43. doi: 10.1093/cvr/cvq318. Epub 2010 Oct 14. PMID 20952413
- [Background] Bastarrika G, Brabham WW, O'Brien TX, Costello P, Schoepf UJ. Dual-source computed tomography assessment of malfunctioning mechanical prosthetic valve. Ann Thorac Surg. 2009 May;87(5):e50. doi: 10.1016/j.athoracsur.2009.02.044. No abstract available. PMID 19379857
- [Background] Jansen AH, Bracke FA, van Dantzig JM, Meijer A, van der Voort PH, Aarnoudse W, van Gelder BM, Peels KH. Correlation of echo-Doppler optimization of atrioventricular delay in cardiac resynchronization therapy with invasive hemodynamics in patients with heart failure secondary to ischemic or idiopathic dilated cardiomyopathy. Am J Cardiol. 2006 Feb 15;97(4):552-7. doi: 10.1016/j.amjcard.2005.08.076. Epub 2006 Jan 4. PMID 16461055
- [Background] Shinbane JS, Chu E, DeMarco T, Sobol Y, Fitzpatrick AP, Lau DM, Klinski C, Schiller NB, Griffin JC, Chatterjee K. Evaluation of acute dual-chamber pacing with a range of atrioventricular delays on cardiac performance in refractory heart failure. J Am Coll Cardiol. 1997 Nov 1;30(5):1295-300. doi: 10.1016/s0735-1097(97)00307-0. PMID 9350930
- [Background] Hochleitner M, Hortnagl H, Hortnagl H, Fridrich L, Gschnitzer F. Long-term efficacy of physiologic dual-chamber pacing in the treatment of end-stage idiopathic dilated cardiomyopathy. Am J Cardiol. 1992 Nov 15;70(15):1320-5. doi: 10.1016/0002-9149(92)90769-u. PMID 1442585
- [Background] Guardigli G, Ansani L, Percoco GF, Toselli T, Spisani P, Braggion G, Antonioli GE. AV delay optimization and management of DDD paced patients with dilated cardiomyopathy. Pacing Clin Electrophysiol. 1994 Nov;17(11 Pt 2):1984-8. doi: 10.1111/j.1540-8159.1994.tb03785.x. PMID 7845803
- [Background] Auricchio A, Salo RW. Acute hemodynamic improvement by pacing in patients with severe congestive heart failure. Pacing Clin Electrophysiol. 1997 Feb;20(2 Pt 1):313-24. doi: 10.1111/j.1540-8159.1997.tb06176.x. PMID 9058869
- [Background] Gill RM, Jones BD, Corbly AK, Ohad DG, Smith GD, Sandusky GE, Christe ME, Wang J, Shen W. Exhaustion of the Frank-Starling mechanism in conscious dogs with heart failure induced by chronic coronary microembolization. Life Sci. 2006 Jul 4;79(6):536-44. doi: 10.1016/j.lfs.2006.01.045. Epub 2006 Apr 19. PMID 16624328
- [Background] Holubarsch C, Ruf T, Goldstein DJ, Ashton RC, Nickl W, Pieske B, Pioch K, Ludemann J, Wiesner S, Hasenfuss G, Posival H, Just H, Burkhoff D. Existence of the Frank-Starling mechanism in the failing human heart. Investigations on the organ, tissue, and sarcomere levels. Circulation. 1996 Aug 15;94(4):683-9. doi: 10.1161/01.cir.94.4.683. PMID 8772688
- [Background] Weil J, Eschenhagen T, Hirt S, Magnussen O, Mittmann C, Remmers U, Scholz H. Preserved Frank-Starling mechanism in human end stage heart failure. Cardiovasc Res. 1998 Feb;37(2):541-8. doi: 10.1016/s0008-6363(97)00227-7. PMID 9614508
- [Background] Schwinger RH, Bohm M, Koch A, Schmidt U, Morano I, Eissner HJ, Uberfuhr P, Reichart B, Erdmann E. The failing human heart is unable to use the Frank-Starling mechanism. Circ Res. 1994 May;74(5):959-69. doi: 10.1161/01.res.74.5.959. PMID 8156643
- [Background] De Vecchis R, Ariano C. Conversion to and maintenance of sinus rhythm do not yield a significant increase in stroke-volume in HFREF patients, whose heart works on the flat branch of Frank-Starling curve, thereby making the retrieval of the atrial mechanical contribution in this subset a substantially futile choice. Eur Heart J. 2019 Nov 21;40(44):3651-3652. doi: 10.1093/eurheartj/ehz655. No abstract available. PMID 31750524
- [Background] Starling EH, Visscher MB. The regulation of the energy output of the heart. J Physiol. 1927 Jan 12;62(3):243-61. doi: 10.1113/jphysiol.1927.sp002355. No abstract available. PMID 16993846
- [Background] Wong JA, Yee R, Stirrat J, Scholl D, Krahn AD, Gula LJ, Skanes AC, Leong-Sit P, Klein GJ, McCarty D, Fine N, Goela A, Islam A, Thompson T, Drangova M, White JA. Influence of pacing site characteristics on response to cardiac resynchronization therapy. Circ Cardiovasc Imaging. 2013 Jul;6(4):542-50. doi: 10.1161/CIRCIMAGING.111.000146. Epub 2013 Jun 5. PMID 23741053
- [Background] Leyva F, Foley PW, Chalil S, Ratib K, Smith RE, Prinzen F, Auricchio A. Cardiac resynchronization therapy guided by late gadolinium-enhancement cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2011 Jun 13;13(1):29. doi: 10.1186/1532-429X-13-29. PMID 21668964
- [Background] Chalil S, Foley PW, Muyhaldeen SA, Patel KC, Yousef ZR, Smith RE, Frenneaux MP, Leyva F. Late gadolinium enhancement-cardiovascular magnetic resonance as a predictor of response to cardiac resynchronization therapy in patients with ischaemic cardiomyopathy. Europace. 2007 Nov;9(11):1031-7. doi: 10.1093/europace/eum133. Epub 2007 Oct 12. PMID 17933857
- [Background] Bleeker GB, Schalij MJ, Van Der Wall EE, Bax JJ. Postero-lateral scar tissue resulting in non-response to cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2006 Aug;17(8):899-901. doi: 10.1111/j.1540-8167.2006.00499.x. PMID 16903969
- [Background] Wouters PC, van Everdingen WM, Vernooy K, Geelhoed B, Allaart CP, Rienstra M, Maass AH, Vos MA, Prinzen FW, Meine M, Cramer MJ. Does mechanical dyssynchrony in addition to QRS area ensure sustained response to cardiac resynchronization therapy? Eur Heart J Cardiovasc Imaging. 2022 Nov 17;23(12):1628-1635. doi: 10.1093/ehjci/jeab264. PMID 34871385
- [Background] Young JB, Abraham WT, Smith AL, Leon AR, Lieberman R, Wilkoff B, Canby RC, Schroeder JS, Liem LB, Hall S, Wheelan K; Multicenter InSync ICD Randomized Clinical Evaluation (MIRACLE ICD) Trial Investigators. Combined cardiac resynchronization and implantable cardioversion defibrillation in advanced chronic heart failure: the MIRACLE ICD Trial. JAMA. 2003 May 28;289(20):2685-94. doi: 10.1001/jama.289.20.2685. PMID 12771115
- [Background] McAlister FA, Ezekowitz J, Hooton N, Vandermeer B, Spooner C, Dryden DM, Page RL, Hlatky MA, Rowe BH. Cardiac resynchronization therapy for patients with left ventricular systolic dysfunction: a systematic review. JAMA. 2007 Jun 13;297(22):2502-14. doi: 10.1001/jama.297.22.2502. PMID 17565085
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430